CLINICAL TRIAL: NCT01411631
Title: A Study to Investigate the Effect of Concord Grape Juice on Cognitive Function in Mums of Preteen Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Welch's, Inc. (Industry)
Responsible Party: Principal Investigator, Prof Louise Dye, Professor, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11-0026
Record Dates: First submitted 2011-06-07; First posted 2011-08-08 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Cognition
Keywords: Polyphenols; Cognition; Cognitive function; Driving performance; Stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grape juice (Active Comparator): Participants will drink 100% concord grape juice daily for 12 weeks
  Interventions: Dietary Supplement: Grape juice polyphenols
- Placebo drink (Placebo Comparator): Participants will drink the placebo for 12 weeks. The placebo will be equicaloric and matched on appearance, taste, volume and macronutrient composition to the grape juice drink.
  Interventions: Dietary Supplement: Grape juice polyphenols

INTERVENTIONS:
Dietary Supplement: Grape juice polyphenols — Participants will consume grape juice polyphenols for 12 weeks and a control juice for 12 weeks.

SUMMARY:
There is some evidence that polyphenols can affect cognitive function. Therefore, consumption of polyphenols has the potential to prevent cognitive impairment or even enhance cognitive performance. The objective of this study is to investigate the effect of polyphenol consumption served in the form of Concord Grape Juice (CGJ) on cognitive performance and driving performance in Mums.

The study design will be a repeated measures, double-blind, randomised, placebo controlled, crossover study. There will be 2 conditions; CGJ and a placebo drink. 20 participants will undergo two 12 week dietary interventions which will entail daily consumption of a 12oz serving of CGJ or placebo in a counterbalanced manner. There will be a 4 week washout period between conditions. At baseline, 6, and 12 weeks of each 12-week treatment arm cognitive performance and driving performance will be assessed (using the driving simulator at the Institute for Transport Studies). CGJ is a common ingredient in commercially available products.

Mums will be defined as mothers of pre-teen children (aged under 13 years) who are aged 40-50. This population generally have hectic and stressful lifestyles and therefore there is potential for this population to receive cognitive benefit from polyphenol consumption.

ELIGIBILITY:
Inclusion Criteria:

* BMI within normal/overweight range (18 - 29 kg/m2)
* Non-smokers or given up more than 6 months ago
* Working 80% of a full time week (at least 30 hours/week)
* Ability to adequately understand verbal and written information in English
* Full Driving Licence held for at least 5 years
* Mothers of pre-teen children (must have child aged <13 years)
* Willing to abstain from drinking red wine and dark fruit juices (e.g. other grape juices, cranberry, raspberry and pomegranate juices) during the study

Exclusion Criteria:

* Menopausal
* diabetes or known impaired glucose tolerance
* taking any regular medication e.g. for hypertension
* Food allergies to ingredients and food colouring of the drinks to be consumed within the study
* Night shift work
* Pregnant or planning a pregnancy within the next year
* Having been pregnant or lactating within the previous 6 months
* Vegetarian
* No history of, or current eating disorders
* Epilepsy (driving SIM exclusion criterion)
* Claustrophobia (driving SIM exclusion criterion)

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive function & Driving Performance | Measured at baseline, baseline+6 weeks, and baseline+12 weeks of each experimental arm
  Cogntive function will be assessed with a battery of cognitive tests, including tests of memory, problem solving skills, concentration, and attention. Driving performance will be assessed using a driving simulator.

SECONDARY OUTCOMES:
Blood Pressure | Measured at baseline, baseline+6 weeks, and baseline+12 weeks of each experimental arm
  Blood pressure measures will be taken over a period before, during and after the driving tasks using an ambulatory blood pressure monitor. An Omron M7 ambulatory blood pressure monitor will be used and can be worn during the driving task.
Subjective Stress | Measured at baseline, baseline+6 weeks, and baseline+12 weeks of each experimental arm
  The sample will be characterised in terms of their psychological stress using the Perceived Stress Scale (PSS, Cohen et al., 1983) the Cook-Medley Hostility Scale (Cook & Medley, 1954), and the Spielberger STAI (Spielberger, 1983) administeredat screening. The PSS and the Spielberger MSTAI will also be administered on each test day.
Subjective ratings of appetite, mood, mental alertness, and concentration | Measured at baseline, baseline+6 weeks, and baseline+12 weeks of each experimental arm
  Measured using visual analogue scales a regular intervals throughout the test day.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Dye, PhD (Professor), Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Institute of Psychological Sciences, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Lamport DJ, Lawton CL, Merat N, Jamson H, Myrissa K, Hofman D, Chadwick HK, Quadt F, Wightman JD, Dye L. Concord grape juice, cognitive function, and driving performance: a 12-wk, placebo-controlled, randomized crossover trial in mothers of preteen children. Am J Clin Nutr. 2016 Mar;103(3):775-83. doi: 10.3945/ajcn.115.114553. Epub 2016 Feb 10. PMID 26864371